CLINICAL TRIAL: NCT06869460
Title: STEREOMIC: Studio Retrospettivo Multicentrico Su Pazienti Trattati Con Radiochirurgia/Radioterapia STEREotassica Per Lesioni Encefaliche Singole. Valutazione Di Efficacy E Safety Del Trattamento Anche Mediante Metodiche Di Analisi RadiOMICa
Brief Title: Multicenter Retrospective Study on Patients Treated with Stereotactic Radiosurgery/Radiotherapy for Single Brain Lesions: Evaluation of Treatment Efficacy and Safety, Also Through Radiomic Analysis Methods.
Acronym: STEREOMIC
Status: Active, not recruiting | Type: Observational
Sponsor: Gemelli Molise Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CET20-02-2024
Record Dates: First submitted 2025-02-20; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Brain Metastases; Radiotherapy Side Effect
Keywords: Brain metastases; Radiotherapy; Stereotactic Body Radiotherapy; Radiosurgery; Radionecrosis; Local Control; Safety profile; Radiomics
MeSH Terms: conditions — Brain Neoplasms; Radiation Injuries | interventions — Radiosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with a singular brain metastases: The study design concerns all patients diagnosed with brain metastases who underwent stereotactic radiosurgery/radiotherapy between January 2010 and December 2022
  Interventions: Radiation: Stereotactic Body Radiotherapy/Radiosurgery

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy/Radiosurgery — Stereotactic Body Radiotherapy/Radiosurgery
  Other Names: SBRT/SRS

SUMMARY:
The study design concerns all patients diagnosed witha singular brain metastasis who underwent stereotactic radiosurgery/radiotherapy between January 2010 and December 2022

DETAILED DESCRIPTION:
The study will include patients of both sexes diagnosed with single brain metastases who underwent radiosurgical/stereotactic treatment. Attention will be paid to data related to local control, potential recurrence, and/or radionecrosis. Once a sufficient number of treated patients is reached, the feasibility of a radiomic feature analysis will be assessed in order to identify potential correlations and/or predictive values for treatment response or radionecrosis. If the sample size is adequate, participating centers will be asked to share pre- and post-RT MRI (brain MRI with contrast using thin slices) and treatment volumes for radiomic evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Treatment with SRS/SRT techniques for a single secondary brain lesion
* Availability of pre-RT brain MRI with contrast (1mm slice thickness)
* Availability of CT simulation imaging for treatment
* Availability of relevant clinical data in the medical record for the study's objectives
* Follow-up of at least 6 months after the completion of SRS or SRT
* Follow-up evaluation through brain MRI

Exclusion Criteria:

* Age under 18 years
* Lack of clinical/radiological data for the patient
* Unavailability of the required imaging
* Previous whole-brain radiotherapy treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study design concerns all patients diagnosed with brain metastases who underwent stereotactic radiosurgery/radiotherapy between January 2010 and December 2022.
Sampling Method: Non-Probability Sample
Enrollment: 372 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Toxicity profile | due to the retrospective nature of the study, we did not have specific time points.We will evaluate the possible onset of toxicity events from the last day of treatment up to 18 months from the treatment
  "The toxicity profile of the treatment will be assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) of the National Cancer Institute."
Local control | We will evaluate Lc at one, two, and five years from the treatment
  It will be Calculated 'per lesion,' and it is defined as the time interval between irradiation and the onset of disease recurrence at the site of the treated area

CONTACTS AND LOCATIONS:
Overall Officials: Donato Pezzulla, M.D., Principal Investigator — Responsible Research Hospital
Locations (4):
- Italy (4):
  - Presidio Ospedaliero "S. G. Moscati", Taranto, Apulia
  - INT IRCCS Fondazione G. Pascale Napoli, Napoli, Campania
  - IRCCS Ospedale San Raffaele, Milan, Lombardy
  - Responsible Research Hospital, Campobasso, Molise